CLINICAL TRIAL: NCT03712501
Title: Influence of Prior Walking on Postprandial Metabolism and Endothelial Function in South Asian vs White European Women.
Brief Title: Influence of Prior Walking on Postprandial Metabolism and Endothelial Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Matthew Roberts, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R16-P188
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases; Endothelial Dysfunction; Insulin Resistance; Oxidative Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants will walk for 60 minutes at 60% maximal oxygen uptake on day 1. Participants will return the following day and consume a high fat breakfast and lunch.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Participants will rest on day 1. Participants will return the following day where they will consume a high fat breakfast and lunch.

INTERVENTIONS:
Behavioral: Exercise — A 60 minute walk at 60% maximal oxygen uptake.
  Arms: Exercise

SUMMARY:
The present study will investigate the effect of prior walking on postprandial metabolism and endothelial function in healthy South Asian and White European women.

Participants will complete two, 2-day trials in a random, crossover design separated by at least 3 weeks to control for the menstrual cycle phase.

On day 1, participants will either rest or complete a 60 minute walk at 60% maximal oxygen uptake. On day 2, participants will arrive at 08:00 having fasted overnight and a baseline venous blood sample and endothelial function measurement will be taken. Participants will consume a high-fat breakfast and lunch and 12 subsequent venous blood samples will be taken throughout the day at standardised intervals to measure a variety of coronary heart disease risk markers. A second endothelial function measurement will be completed 2 hours after the breakfast. Blood pressure will be measured every hour.

It is expected that the South Asian participants will have impaired metabolism and endothelial function compared to their European counterparts but the bout of exercise performed on day 1 will mitigate these responses.

DETAILED DESCRIPTION:
South Asian individuals have a higher-than-average risk of coronary heart disease. The reasons for this are unclear, but physical inactivity and/or poor responsiveness to exercise may play a role.

Previous research from our laboratory has shown that coronary heart disease risk markers in the postprandial period are elevated in South Asian men, but acute exercise was equally, if not more, effective for reducing these risk markers in South Asian than White European men. However, the effect of acute exercise on coronary heart disease risk markers has not been examined in South Asian women.

Therefore, the purpose of the present study is to compare the effect of acute exercise on endothelial function and coronary heart disease risk markers in women of South Asian versus White European descent.

On visit 1, participants will attend the laboratory to undergo preliminary assessments and to be familiarised with the laboratory environment and study procedures. Specifically, health status, habitual physical activity, dietary habits and anthropometric data (height, weight, waist and hip circumference, body fat) will be collected. Two preliminary exercise tests will be performed as follows: 1) submaximal-incremental treadmill walking test and 2) incremental treadmill running test to exhaustion to measure maximal oxygen uptake.

On visit 2, participants will undergo a magnetic resonance imaging (MRI) scan to quantify regional body composition comprising abdominal subcutaneous adipose tissue, visceral adipose tissue, liver fat percentage, thigh intramuscular adipose tissue and thigh muscle volume.

On visits 3-6 participants will complete two, 2-day trials in a random, crossover design seperated by at least 3 weeks to control for the menstrual cycle phase. On day 1 of both trials, participants will arrive fasted at 08:00 and a baseline blood sample, blood pressure and endothelial function measurement will be taken. Participants will consume a standardised high fat breakfast at 09:00 and lunch at 13:00. At 15:30 the participants will walk for 60 minutes at 60% maximal oxygen uptake and complete a second endothelial function measurement at 16:45. Participants will leave the laboratory with a standardised evening meal to consume before 22:00. The control trial will be the same, except no exercise will be performed.

On day 2, participants will arrive at 08:00 having fasted overnight for 10h (except plain water). A cannula will be inserted into the antecubital vein for collection of venous blood samples. Blood pressure will be measured at 08:00 (0h) and again at hourly intervals throughout the day. Endothelial function will measured at 08:15 (0.25h) and again at 3h. At 0h, a fasting blood sample will be collected. Subsequent venous blood samples will be collected at 1.5, 1.75, 2, 3, 4, 5, 5.5, 5.75, 6, 7, 8 and 9h. Participants will consume a standardised high fat breakfast at 1h and a standardised high fat lunch at 5h. The meals consist of 57% fat, 32% carbohydrate and 11% protein. The meals provide 14.3 kcal per kg of body mass.

Participants will rest in the laboratory throughout day 2 of both the exercise and control trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 year old South Asian and White European women;
* Be able to walk continuously for 1 hour;
* Weight stable for the past 3 months;
* Non-smokers;
* No known contradictions to maximal exertion exercise (e.g., recent musculoskeletal injury, congenital heart disease).

Exclusion Criteria:

* Musculoskeletal injury that has affected normal ambulation within the last month;
* Congenital heart disease;
* Any muscle or bone injuries that do not allow them to walk on a treadmill;
* Uncontrolled exercise-induced asthma;
* Coagulation or bleeding disorders;
* Diabetes (metabolism will be different to non-diabetics potentially skewing the data);
* Taking any medication that might influence fat metabolism;
* Taking any medication that might influence blood glucose (e.g., insulin for diabetes);
* Heart conditions;
* Smoking;
* Dieting or restrained eating behaviours;
* Weight fluctuation greater than 3 kg in the previous 3 months to study enrolment;
* A food allergy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Triacylglycerol | Day 1 fasting. Day 2 fasting, 1.5h, 1.75h, 2h, 3h, 4h, 5h, 5.5h, 5.75h, 6h, 7h, 8h and 9h.
  Fasting on day 1 and 2. Time-course of plasma triacylglycerol concentrations in response to exercise and/or feeding on day 2.

SECONDARY OUTCOMES:
Endothelial function | Day 1 fasting and 8.75h. Day 2 fasting and 3.5h.
  Changes in endothelial function via flow-mediated dilatation in response to feeding and exercise.
Blood pressure | Day 1 fasting. Day 2 fasting and 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h and 9h.
  Changes in blood pressure (systolic and diastolic).
Glucose | Day 1 fasting. Day 2 fasting, 1.5h, 1.75h, 2h, 3h, 4h, 5h, 5.5h, 5.75h, 6h, 7h, 8h and 9h
  Fasting on day 1 and 2. Time-course of plasma glucose concentrations in response to exercise and/or feeding on day 2.
Total cholesterol | Day 1 fasting. Day 2 fasting.
  Fasting plasma total cholesterol on day 1 and day 2 of both trials.
Insulin | Day 1 fasting. Day 2 fasting, 1.5h, 2h, 4h, 5h, 5.5h, 7h, 8h.
  Fasting on day 1 and 2. Time-course of plasma insulin concentrations in response to exercise and/or feeding on day 2.
High-density lipoprotein cholesterol | Day 1 fasting. Day 2 fasting.
  Fasting high-density lipoprotein cholesterol on day 1 and 2 of both trials.
Low-density lipoprotein cholesterol | Day 1 fasting. Day 2 fasting.
  Fasting low-density lipoprotein cholesterol on day 1 and 2 of both trials.
Non-esterified fatty acids | Day 1 fasting. Day 2 fasting, 1.5h, 2h, 4h, 5h, 5.5h, 7h and 9h.
  Fasting on day 1 and 2. Time-course of plasma non-esterified fatty acid concentrations in response to exercise and/or feeding on day 2.
Interleukin-6 | Day 1 fasting. Day 2 fasting, 3h, 6h and 8h.
  Fasting on day 1 and 2. Time-course of plasma interleukin-6 concentrations in response to exercise and/or feeding on day 2.
C-Reactive protein | Day 1 fasting. Day 2 fasting, 3h, 6h and 8h.
  Fasting on day 1 and 2. Time-course of plasma C-Reactive protein concentrations in response to exercise and/or feeding on day 2.
Peroxiredoxin-4 | Day 1 fasting. Day 2 fasting, 3h, 6h and 8h.
  Fasting on day 1 and 2. Time-course of plasma peroxiredoxin-4 concentrations across day 2 of both trials.
Superoxide dismutase 3 | Day 1 fasting. Day 2 fasting, 3h, 6h and 8h.
  Fasting on day 1 and 2. Time-course of plasma Superoxide dismutase 3 concentrations across day 2 of both trials

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Roberts, Principal Investigator — Loughborough University
Locations (1):
- National Centre for Sport and Exercise Medicine, Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised individual participant data for all primary and secondary outcome measures will be made available.

REFERENCES:
- [Background] Arjunan SP, Deighton K, Bishop NC, King J, Reischak-Oliveira A, Rogan A, Sedgwick M, Thackray AE, Webb D, Stensel DJ. The effect of prior walking on coronary heart disease risk markers in South Asian and European men. Eur J Appl Physiol. 2015 Dec;115(12):2641-51. doi: 10.1007/s00421-015-3269-7. Epub 2015 Oct 5. PMID 26438068
- [Background] Arjunan SP, Bishop NC, Reischak-Oliveira A, Stensel DJ. Exercise and coronary heart disease risk markers in South Asian and European men. Med Sci Sports Exerc. 2013 Jul;45(7):1261-8. doi: 10.1249/MSS.0b013e3182853ecf. PMID 23470315
- [Derived] Roberts MJ, Thackray AE, Wadley AJ, Alotaibi TF, Hunter DJ, Thompson J, Fujihira K, Miyashita M, Mastana S, Bishop NC, O'Donnell E, Davies MJ, King JA, Yates T, Webb D, Stensel DJ. Effect of Acute Walking on Endothelial Function and Postprandial Lipemia in South Asians and White Europeans. Med Sci Sports Exerc. 2023 May 1;55(5):794-802. doi: 10.1249/MSS.0000000000003098. Epub 2022 Dec 5. PMID 36729923

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03712501/SAP_000.pdf